CLINICAL TRIAL: NCT00085176
Title: Neurobehavioral Outcomes in Childhood Acute Lymphoblastic Leukemia. A Limited Non-Therapeutic Study
Brief Title: Neurobehavioral Complications in Children Who Were Previously Treated With Steroids and Intrathecal Therapy for Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ALTE02C2; COG-ALTE02C2 (Other: Children's Oncology Group); CDR0000367480 (Other: Clinicaltrials.gov)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Leukemia; Long-term Effects Secondary to Cancer Therapy in Children; Neurotoxicity; Psychosocial Effects of Cancer and Its Treatment
Keywords: long-term effects secondary to cancer therapy in children; neurotoxicity; psychosocial effects of cancer and its treatment; childhood acute lymphoblastic leukemia in remission
MeSH Terms: conditions — Leukemia; Neurotoxicity Syndromes | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: management of therapy complications
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Cancer therapies may affect the ability of a child's brain and central nervous system to function normally. Learning to identify which patients will develop complications may improve the ability of doctors to plan cancer treatment and improve patient quality of life.

PURPOSE: This clinical trial is studying neurobehavioral changes in children who have received steroid therapy or intrathecal therapy for acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare neurobehavioral functioning, specifically memory, attention, executive function, visual-motor integration, and processing speed, in children previously treated with steroids (prednisone vs dexamethasone) and intrathecal therapy (methotrexate alone vs methotrexate, cytarabine, and hydrocortisone) for childhood acute lymphoblastic leukemia.
* Correlate non-treatment risk factors, such as gender, age at diagnosis, and time since termination of prior therapy, with impaired neurobehavioral function in these patients.
* Correlate neurobehavioral complications with quality-of-life of these patients.

OUTLINE: This is a multicenter, cohort study. Patients are assigned to 1 of 2 cohorts (prior treatment per CCG-1922 [prednisone vs dexamethasone] vs prior treatment per CCG-1952 [intrathecal (IT) methotrexate vs IT methotrexate, cytarabine, and hydrocortisone]). Patients in each cohort are stratified according to age at diagnosis, gender, and time since prior treatment termination.

* Cohort A (CCG-1922): Patients undergo physical and neurological examination, neurobehavioral evaluation, and quality of life assessment. Neurobehavioral evaluations assess memory, attention, and executive function.
* Cohort B (CCG-1952): Patients undergo evaluation as above. Neurobehavioral evaluations assess visual-motor integration and processing speed.

PROJECTED ACCRUAL: A total of 448 patients (224 per cohort) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of standard-risk childhood acute lymphoblastic leukemia (ALL)

  * In continuous first remission
  * No history of CNS pathology requiring radiotherapy or surgery
* Prior enrollment on one of the following Children's Cancer Group (CCG) protocols AND terminated therapy at least 1 year ago:

  * CCG-1922 (prednisone vs dexamethasone)
  * CCG-1952 (intrathecal methotrexate vs triple intrathecal therapy)

    * No prior enrollment on CCG-1952 arm III
* No history of pre-existing neurodevelopmental disorder before diagnosis of ALL (e.g., mental retardation, Down syndrome, seizure disorder, or traumatic brain injury)
* No neuropsychological assessment within the past 6 months

PATIENT CHARACTERISTICS:

Age

* 6.5 to 16 years

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Reading, speaking, and listening comprehension of English by patient required (English and/or Spanish by parent)
* No history of very low birth weight (< 1,500 grams)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics

Other

* Concurrent stimulants allowed

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children previously randomized to (1) dexamethasone instead of prednisone on COG 1922 and (2) intrathecal methotrexate, cytarabine, and hydrocortisone (triple therapy) instead of intrathecal methotrexate alone on COG 1952
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2004-05; Primary Completion 2009-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Two-sided comparisons of various mean neurobehavioral scores between the two treatment arms within each study | length of study
  Data analysis for each of the two clinical trials will be conducted separately. The primary objectives will be two-sided comparisons of various mean neurobehavioral scores between the two treatment arms within each study.

CONTACTS AND LOCATIONS:
Overall Officials: Nina S. Kadan-Lottick, MD, MSPH, Study Chair — Yale University; Joseph P. Neglia, MD, MPH, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (31):
- United States (31):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University Cancer Institute, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

REFERENCES:
- [Result] Lindemulder SJ, Stork LC, Bostrom BC, et al.: Trends in body mass index (BMI) during and after treatment for standard risk (SR) acute lymphoblastic leukemia (ALL): A report from the Children's Oncology Group (COG). [Abstract] J Clin Oncol 30 (Suppl 15): A-9546, 2012.
- [Result] Kadan-Lottick NS, Brouwers P, Breiger D, Kaleita T, Dziura J, Liu H, Chen L, Nicoletti M, Stork L, Bostrom B, Neglia JP. A comparison of neurocognitive functioning in children previously randomized to dexamethasone or prednisone in the treatment of childhood acute lymphoblastic leukemia. Blood. 2009 Aug 27;114(9):1746-52. doi: 10.1182/blood-2008-12-186502. Epub 2009 Jun 22. PMID 19546477
- [Result] Breiger D, Kaleita TA, Kadan-Lottick NS, et al.: Behavioral social adjustment in survivors of childhood acute lymphoblastic leukemia (ALL) treated without cranial radiation. [Abstract] Pediatr Blood Cancer 46 (6): A-3505.43, 690, 2006.
- [Result] Kadan-Lottick NS, Brouwers P, Kaleita TA, et al.: Preliminary findings of neurobehavioral outcomes in survivors of childhood acute lymphoblastic leukemia (ALL) treated without cranial radiation. [Abstract] Pediatr Blood Cancer 46 (6): A-3505.45, 691, 2006.
- [Result] Kadan-Lottick NS, Stork LC, Bostrom BC, et al.: Increased prevalence of overweight status in survivors of acute lymphoblastic leukemia (ALL) treated without cranial radiation . [Abstract] Pediatr Blood Cancer 46 (6): A-3505.44, 690, 2006.